CLINICAL TRIAL: NCT05381168
Title: Efficacy and Safety of Calcium From Fish Bone in Volunteers With Osteopenia
Brief Title: Calcium From Fish Bone in Volunteers With Osteopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 176/64
Record Dates: First submitted 2022-05-05; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Osteopenia
Keywords: osteopenia; calcium; fish bone; efficacy; safety
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Calcium Carbonate

STUDY DESIGN:
Intervention Model Description: The volunteers are divided into 2 groups which are calcium from fish bone treatment group and calcium carbonate treatment group. Both groups receive the calciums every day for 6 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcium from fish bone (Experimental): The volunteer will receive calcium from fish bone 4 capsules per day for 6 months.
  Interventions: Dietary Supplement: Calcium from fish bone
- Calcium carbonate (Active Comparator): The volunteer will receive calcium carbonate 2 tablets per day for 6 months.
  Interventions: Dietary Supplement: Calcium carbonate

INTERVENTIONS:
Dietary Supplement: Calcium from fish bone — Calcium from fish bone contained calcium 312 mg and vitamin D 100 IU per capsule.
  Arms: Calcium from fish bone
Dietary Supplement: Calcium carbonate — Calcium carbonate contained calcium 600 mg and vitamin D 200 IU per capsule.
  Arms: Calcium carbonate

SUMMARY:
The aims of this study are to explore efficacy and safety of calcium from fish bone in volunteers with osteopenia. The volunteers are divided into 2 groups which are calcium from fish bone treatment group and calcium carbonate treatment group. Both groups received the calciums everyday for 6 months. Bone mineral density, blood examination, physical examination, adverse events, and satisfaction are evaluated before and after treatment.

DETAILED DESCRIPTION:
The aims of this study are to explore efficacy and safety of calcium from fish bone in volunteers with osteopenia. The volunteers are divided into 2 groups which are calcium from fish bone treatment group and calcium carbonate treatment group. Both groups received the calciums everyday for 6 months. Bone mineral density is analyzed before and after treatment. Osteocalcin, total procollagen type-1 N-terminal propeptide (P1NP), beta-crosslaps, parathyroid hormone (PTH), calcium, phosphate level, vitamin D level (Serum 25(OH)D), albumin, aspartate transaminase (AST), alanine transaminase (ALT), alkaline phosphatase (ALP), creatinine (Cr), blood urea nitrogen (BUN), and complete blood count (CBC) are assessed before and after taking for 3 and 6 months. Physical performance and food diary are also tested and records. Moreover, adverse effects including skin allergy, gastrointestinal abnormality, respiratory abnormality are evaluated. Satisfaction is asked after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male age more than 70 years or female age more than 65 years or all age volunteers that have at least 1 risk factors which are menopause before 45 years, menopause with the height reduction (more than 4 cm), body mass index less than 20 kg/mm2, bone fracture history, taking some medicine that has an effect on bone density reduction, have disease that has an effect on bone density reduction, Father and mother have bone fracture history, fracture risk assessment tool (FRAX) in intermediate risk, osteoporosis self-assessment tool for asian (OSTA) score, khon kaen osteoporosis study (KKOS) score in intermediate risk or higher intermediate risk
* Bone mineral density between -1 to -2.5
* No osteosclerosis
* Can read and write
* Willing to be volunteer

Exclusion Criteria:

* Allergic to calcium, magnesium, phosphorus, zinc, collagen, and osteocalcin
* Taking calcium or vitamin D with in 14 days before the study start
* Taking osteosclerosis' medicine
* Have uncontrolled diseases
* Pregnancy and lactation
* Participating in other study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-05-20 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density score | 6 months
  Bone mineral density score is measured using dual energy x-ray absorptiometry scanner (DEXA scanner). It shows in term of T-score. The outcomes are compared bone mineral density score of calcium from fish bone group to calcium carbonate group.

SECONDARY OUTCOMES:
Osteocalcin level | 6 months
  Changing of osteocalcin level of calcium from fish bone group compared to calcium carbonate group.
Total procollagen type-1 N-terminal propeptide (P1NP) level | 6 months
  Changing of P1NP level of calcium from fish bone group compared to calcium carbonate group.
Beta-crosslaps level | 6 months
  Changing of beta-crosslaps level of calcium from fish bone group compared to calcium carbonate group.
Parathyroid hormone (PTH) level | 6 months
  Changing of PTH level of calcium from fish bone group compared to calcium carbonate group.
Blood calcium level | 6 months
  Changing of blood calcium level of calcium from fish bone group compared to calcium carbonate group.
Blood phosphate level | 6 months
  Changing of blood phosphate level of calcium from fish bone group compared to calcium carbonate group.
Vitamin D level | 6 months
  Changing of vitamin D level of calcium from fish bone group compared to calcium carbonate group.
Liver function level | 6 months
  Changing of liver function level (aspartate transaminase (AST), alanine transaminase (ALT), alkaline phosphatase (ALP)) of calcium from fish bone group compared to calcium carbonate group.
Creatinine level | 6 months
  Changing of creatinine (Cr) level of calcium from fish bone group compared to calcium carbonate group.
Blood urea nitrogen level | 6 months
  Changing of blood urea nitrogen (BUN) of calcium from fish bone group compared to calcium carbonate group.
Pain score | 6 months
  Changing of pain score using visual analogue scale (0 painless to 10 very pain) of calcium from fish bone group compared to calcium carbonate group.
Short physical performance battery score | 6 months
  Changing of short physical performance battery score (0 weak to 12 very strong)of calcium from fish bone group compared to calcium carbonate group.
Grip strength | 6 months
  Changing of grip strength (kilogram) of calcium from fish bone group compared to calcium carbonate group.
Skin allergic reactions | 6 months
  The outcome measurements of skin allergic reactions are appearance (have or no have) of rash, edema, bullae, pain, and itching.
Respiratory tract abnormality | 6 months
  The outcome measurements of respiratory tract abnormality are appearance (have or no have) of shortness of breath and asthma.
Gastrointestinal tract abnormality | 6 months
  The outcome measurements of gastrointestinal tract abnormality are appearance (have or no have) of nausea, vomiting, flatulence, constipation, and diarrhea.
Satisfaction level | 6 months
  Satisfaction score (0 unsatisfied to 10 very satisfied)